CLINICAL TRIAL: NCT06405022
Title: Does Sport Specific Brain Endurance Training Enhance Physical and Cognitive Performance in Elite Orienteering Athletes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Public Health, Denmark (Other)
Collaborators: Team Denmark (Other)
Responsible Party: Principal Investigator, Simon Lønbro, Teaching Associate Professor, PhD, Department of Public Health, Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BET in orienteering
Record Dates: First submitted 2021-03-16; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Elite Athletes

STUDY DESIGN:
Intervention Model Description: The study is constructed as a cross-over design (Fig. 1), where participants function as their own control condition. The control condition (the first period) and the intervention (the latter period) consists of a 6 week training period, both leading up to a prioritized international competition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (CON) (Active Comparator): The control condition entails a six-week period. The participant will complete three regular high intensity training per week followed by 20 min of rest
  Interventions: Other: Control
- Brain Endurance Training (BET) (Experimental): The intervention period also entails a 6 week period but with three weekly blocks with a 20 min brain endurance training program following a regular high intensity training session.
  Interventions: Other: Brain Endurance Training

INTERVENTIONS:
Other: Brain Endurance Training — Six week period with three weekly blocks with a 20 min brain endurance training program following a regular HIT session. Before the HIT session questionnaires are completed to measure the motivation for the HIT session and the current state of mood. In between the HIT session and the RCA session, questionnaires are completed to measure the experienced workload of the HIT session, the current state of mood, and the motivation for following the RCA session. Immediately after the RCA session, questionnaires are completed to measure the experienced workload of the RCA session and the current state of mood.
  Arms: Brain Endurance Training (BET)
Other: Control — No intervention
  Arms: Control (CON)

SUMMARY:
The purpose of the study is to measure the effects of a 6 week sport specific BET intervention on physical and cognitive performance parameters in elite orienteering athletes.

DETAILED DESCRIPTION:
The purpose of the study is to measure the effects of a 6 week sport specific BET intervention on physical and cognitive performance parameters in elite orienteering athletes.

The study is constructed as a cross-over design, where participants function as their own control condition. The control condition (the first period) and the intervention (the latter period) consists of a 6 week training period, both leading up to a prioritized international competition. In the control condition participants will train normally leading up to the European Championships. During the intervention period participants will implement 3 sessions per week of a specially designed brain endurance program, leading up to the World Championships. To investigate the effect on all endpoints, physical and cognitive tests are conducted before and after the training periods.

ELIGIBILITY:
Inclusion Criteria:

* Danish National Team Elite Orienteering Runners

Exclusion Criteria:

* Consent withdrawal
* Injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Change in 5000 m run performance (time) | At baseline, after 6 (after CON) and after 12 (after BET) weeks
  Self Paced endurance test (physical test part 1) To measure maximal self-paced endurance performance, a track and field test will be performed. This test is completed on a standard athletic track measuring 400m.
Change in Cognitive performance #1 (score) | At baseline, after 6 (after CON) and after 12 (after BET) weeks
  Change in Inhibition task performance (cognitive test part 1a) This cognitive test consists of the Stroop colour-word task. Participants perform this task on a computer whilst sitting in a quiet and dim lit room. Four words (yellow, blue, green, red) are serially presented on the screen until the participant validates an answer which is followed by a 1,500 ms interval.
Change in Cognitive performance #2 (score) | At baseline, after 6 (after CON) and after 12 (after BET) weeks
  Route Choice Assessment program (RCA) (cognitive test part 1b) Participants perform the RCA on a computer whilst sitting comfortably in a quiet and dim lit room. The RCA program is a specially designed computer program. The program contains approximately 1500 different orienteering legs.

SECONDARY OUTCOMES:
1000 m submaximal running performance | At baseline, after 6 (after CON) and after 12 (after BET) weeks
  Lactate levels during a submaximal 1000 m run is measured to assess physiological stress during the submax test.
Mood change | At baseline, after 6 (after CON) and after 12 (after BET) weeks
  The Brunel Mood Scale (BRUMS) is used to assess mood. This questionnaire, which is based on the Profile of Mood States, contains 24 items (e.g., angry, uncertain, miserable, tired, nervous, energetic) divided into six respective subscales: anger, confusion, depression, fatigue, tension, and vigor. The items are answered on a 5-point Likert scale (0 not at all, 1 a little, 2 moderately, 3 quite a bit, 4 extremely), and each subscale, with four relevant items, can achieve a raw score in the range of 0 to 16 with a higher number indicating a stronger expression. Because of the particular interest in mental fatigue in the present study, we specify that an alteration in the subscales for fatigue and vigor is an indication of mental fatigue.
Subjective workload change | At baseline, after 6 (after CON) and after 12 (after BET) weeks
  The National Aeronautics and Space Administration Task Load Index (NASA-TLX) rating scale is used to assess subjective workload. The NASA-TLX is composed of six subscales: mental demand (How much mental and perceptual activity was required?), physical demand (How much physical activity was required?), temporal demand (How much time pressure did you feel due to the rate or pace at which the task occurred?), performance (How much successful do you think you were in accomplishing the goals of the task set by the experimenter?), effort (How hard did you have to work to accomplish your level of performance?) and frustration (How much irritating or annoying did you perceive the task?). The participants scores on each of the items on a scale divided into 20 equal intervals anchored by a bipolar descriptor (e.g. high/low). This score is multiplied by 5, resulting in a final score between 0 and 100 for each of the subscales with a higher number indicating a higher workload.
Motivation change | At baseline, after 6 (after CON) and after 12 (after BET) weeks
  Motivation is measured using the visual analogue scale (VAS) with 1 item (How motivated do you feel for the upcoming task?) The VAS scale consists of a 100-mm line anchored by a bipolar descriptor (not at all / a lot), on which participants mark their answer. Participants are instructed to answer VAS regarding their feeling of motivation for the upcoming task. The mark is transferred to a final score between 0 and 100 corresponding to the actual physical placement of the mark on the scale. A higher number indicating a high amount of motivation.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: Undecided